CLINICAL TRIAL: NCT05805254
Title: Neurofunctional Study of the Brain Activity of Preterm Infants During Family-centered Interventions
Brief Title: Neurofunctional Study of Preterm Infants' Brain Activity
Status: Completed | Type: Observational
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 02/17
Record Dates: First submitted 2023-03-24; First posted 2023-04-07 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Brain Activity; Preterm
Keywords: Preterm infant; Kangaroo Mother care; family-centered interventions; near-infrared spectroscopy
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During hospital stay, a family centered therapeutic approach is increasingly seen as the preferred clinical and care model to be adopted, since it is effective in promoting the neurobehavioral development of the infant and the psychophysical health of the family. In preterm infant, parental relationship and parental relationship-centered interventions, such as kangaroo mother care (KMC), are actively promoted. Studies carried out with electroencephalography showed that preterm infants who participated in KMC interventions have, when reach term equivalent age, a similar level of maturity as healthy full-term infants. It has also been observed that KMC carried out in preterm infant with gestational age <33 weeks promotes adequate development of the primary motor cortex during adolescence.

Recent scientific evidence showed an early response to relational stimulations, in particular to their emotional content, of term infants. After few days of life, the infant's brain picks up messages from the human context and interacts with them. For example, a study using near-infrared spectroscopy (NIRS) showed increased activation of the right frontal cortex in infants in association with their mother's direct speech. Similar neuroimaging studies have not yet been conducted in preterm infants during hospitalization. The aim of this study is to assess the activation of the cerebral cortex of the preterm infant in the course of 1) KMC and 2) listening to their mother's voice, using optical topography, a multichannel NIRS system.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at birth ≤32 weeks
* absence of brain injury and neurological problems
* newborn-mother pairs in KMC
* adherence to research by parents.

Exclusion Criteria:

* contraindications to KMC and NIRS, according to internal protocol

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants with gestational age at birth ≤32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-03-25 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Values of cortical oxy-haemoglobin (HbO2) during KMC in preterm infants | During hospital stay, between 30 to 36 weeks of postmenstrual age
  Multichannel near-infrared spectroscopy will be used to estimate cerebral cortex activation by measuring cortical oxy-haemoglobin (HbO2) values

SECONDARY OUTCOMES:
Values of cortical oxy-haemoglobin (HbO2) during the experience of listening the mother's voice and the voice of an unknown woman in preterm infants | During hospital stay, between 30 to 36 weeks of postmenstrual age
  Multichannel near-infrared spectroscopy will be used to estimate cerebral cortex activation by measuring cortical oxy-haemoglobin (HbO2) values

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Bembich, MSC, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy